CLINICAL TRIAL: NCT03101735
Title: A Real Life, Non-interventional, Multicentre Study to Assess Resource Utilization and Quality of Life of Patients With Relapsing Forms of Multiple Sclerosis Treated With Dimethyl Fumarate in Greece - the FIDELITY Study
Brief Title: Study to Assess Resource Utilization and Quality of Life of Patients With RRMS Treated With Tecfidera in Greece
Acronym: FIDELITY
Status: Completed | Type: Observational
Sponsor: Genesis Pharma CNS & Specialty (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-GEN-DMF-001
Record Dates: First submitted 2017-03-03; First posted 2017-04-05 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2020-02

CONDITIONS: RRMS
MeSH Terms: interventions — Dimethyl Fumarate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Dimethyl Fumarate (DMF) — The non-interventional design allows the observation of patients in a broad range of settings reflecting routine clinical practice. All decisions on therapeutic or diagnostic procedures, treatments, management of the disease, or resource utilisation will be at the full discretion of the treating physician without interference by a sponsor or study protocol. All treatment decisions will follow the real-life treatment behaviour.
  Other Names: Tecfidera

SUMMARY:
This is a non interventional, multicenter clinical trial, in adult patients receiving Tecfidera per approved SmPC and routine clinical practice. The primary objective of this study is to evaluate the total societal costs to the healthcare system related to the use of Tecfidera in RRMS patients. The study will capture data in a simple matter that can be easily interpreted providing an advantage in a country where efforts in the market access arena are in their infancy. For the aforementioned reasons, the proposed study may prove quite valuable in supporting DMF as a cost-effective therapy, valuable not only for patients but for the public health care system as well, providing all the necessary information for the evaluation that need to be examined regarding the positive reimbursement list and future decisions.

DETAILED DESCRIPTION:
The study will take place in Greece. Investigators will participate from a broad geographical distribution in order to ensure a proper representation from all areas of Greece. Investigator's decision to prescribe DMF (Tecfidera®) (according to the indication for treatment as defined in the summary of product characteristics, SmPC and the current clinical practice), should precede entry into the study.

ELIGIBILITY:
Inclusion Criteria:

* Persons aged 18-65 years.
* Patients with a confirmed diagnosis of RRMS.
* Patients for whom the decision to prescribe therapy with Tecfidera®, according to the locally approved product's summary of product characteristics (SmPC) has already been taken prior to their enrolment in the study. The assignment of a patient to this therapeutic strategy is not decided in advance, but falls within current practice, while the prescription of Tecfidera® is clearly separated from the physician's decision to include the patient in the current study.
* Patients must have signed an informed consent document.
* Patients must be able to read, understand and complete the study specific questionnaire.

Exclusion Criteria:

* Patients having other forms of MS, like Clinically Isolated Syndrome (CIS) or progressive forms.
* Patients who have initiated treatment with Tecfidera® more than 7 days before study enrolment or have received DMF at any different time prior to this period.
* Patients that meet any of the contraindications to the administration of the study drug according to the approved SmPC.
* Receipt of any investigational agent within 30 days or 5 half-lives of the investigational agent (whichever is longer) before the commencement of therapy with Tecfidera®.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 400 previously DMF-naïve adult patients who have been diagnosed with RRMS and will initiate treatment with Dimethyl Fumarate up to 1 week before study enrolment will be included
Sampling Method: Non-Probability Sample
Enrollment: 455 (Actual)
Dates: Start 2016-09-23 (Actual); Primary Completion 2020-04-23 (Actual); Study Completion 2020-04-23 (Actual)

PRIMARY OUTCOMES:
Total Cost | The primary outcome measure will be assessed at 6, 12, 18 and 24 months post recruitment. The data that will be presented is the total societal costs to the healthcare system related to the use of Tecfidera.
  The primary endpoint of this study is the total cost, at the end of the study, of treatment, of the utilization of healthcare services, and of personal expenses associated with RRMS in patients receiving Dimethyl Fumarate.

CONTACTS AND LOCATIONS:
Locations (1):
- University General Hospital AHEPA (B'), Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kourlaba G, Koutsis G, Fakas N, Tsimourtou V, Karachalios G, Bakirtzis C, Grigoriadis N. The economic impact, healthcare resource utilization, and clinical outcome over 24 months in patients with relapsing-remitting multiple sclerosis treated with dimethyl fumarate in Greece- The Fidelity Study. Expert Rev Pharmacoecon Outcomes Res. 2025 Dec 18:1-11. doi: 10.1080/14737167.2025.2603955. Online ahead of print. PMID 41390331